CLINICAL TRIAL: NCT06530914
Title: A Phase II Study of MRG003 Injection Combined With Pucotenlimab Injection ± Cisplatin Injection in the Neoadjuvant Treatment Locally Advanced EGFR-positive Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Liu (Other)
Responsible Party: Sponsor-Investigator, Lei Liu, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-HNC-II-007
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Locally Advanced EGFR-positive HNSCC; Neoadjuvant therapy; Antibody-drug conjugate; immunotherapy; chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG003+Pucotenlimab (Experimental): Neoadjuvant:
  Patients receive MRG003 in combination with Pucotenlimab for 3 cycles before surgery.
  Surgery:
  Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Adjuvant:
  Patients receive adjuvant Pucotenlimab for 8 cycles.
  Interventions: Drug: MRG003 combined with Pucotenlimab
- MRG003+Pucotenlimab+Cisplatin (Experimental): Neoadjuvant:
  Patients receive MRG003 in combination with Pucotenlimab + cisplatin for 3 cycles before surgery.
  Surgery:
  Within a 2-6 week window post induction, tumor imaging will be followed by surgical resection.
  Adjuvant:
  Patients receive adjuvant Pucotenlimab for 8 cycles.
  Interventions: Drug: MRG003 combined with Pucotenlimab+Cisplatin

INTERVENTIONS:
Drug: MRG003 combined with Pucotenlimab — Both interventions all drugs intravenous infusion, D1, once every 3 weeks, a total of 3 cycles.
  Other Names: MRG003+Pucotenlimab
  Arms: MRG003+Pucotenlimab
Drug: MRG003 combined with Pucotenlimab+Cisplatin — All interventions all drugs intravenous infusion, once every 3 weeks, a total of 3 cycles.
  Other Names: MRG003+Pucotenlimab+Cisplatin
  Arms: MRG003+Pucotenlimab+Cisplatin

SUMMARY:
A Randomized, Phase II Study of MRG003 in Combination With Pucotenlimab Injection ± Cisplatin in Patients With Locally Advanced EGFR-positive Head and Neck Squamous Cell Carcinoma. This proposed study will evaluate the efficacy and safety of preoperative administration of MRG003 in Combination With Pucotenlimab Injection ± Cisplatin in HNSCC who are eligible for resection.

DETAILED DESCRIPTION:
In this study, eligible patients will be randomized in a 1:1 ratio to either the MRG003 Injection Combined With Pucotenlimab Injection treatment group (Cohort 1), or the MRG003 Injection Combined With Pucotenlimab Injection + Cisplatin treatment group (Cohort 2). Pathological response rate will be the primary outcome measures. Adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent voluntarily and follow the requirements of the program;
2. Age ≥18 years old, ≤70 years old, gender is not limited;
3. Physical condition score ECOG 0 or 1;
4. Histopathology confirmed the diagnosis of head and neck squamous cell carcinoma, and immunohistochemistry confirmed that EGFR expression was positive (defined as weak staining of > 10% of tumor cells);
5. No previous treatment for head and neck squamous cell carcinoma, including drug therapy, radiotherapy, surgery, etc., and the tumors of the subjects assessed by the researchers before admission could be surgically resected;
6. According to the American Joint Committee on Cancer (AJCC) /TNM Staging System eighth Edition, patients must have the following tumor stages: 1) patients with stage III, IVA, and IVB non-oropharyngeal cancer and patients with HPV-negative oropharyngeal cancer; Or 2) Stage II and III HPV-positive oropharyngeal cancer patients. For patients with oropharyngeal cancer, HPV status should be determined by p16 IHC.
7. The level of organ function must meet the following requirements:

   * Bone marrow: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L, and no blood transfusion or biological response regulator (such as granulocyte, erythrocyte growth factor, etc.) treatment within 14 days before the first dose;
   * Liver: total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤2.5×ULN; Serum albumin ≥28 g/L;
   * Kidney: creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula);
   * Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5×ULN (except those receiving therapeutic anticoagulants);
   * No severe cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%;
8. Fertile men and women of childbearing age are willing to take effective contraceptive measures from the signing of informed consent to 6 months after the last administration of the experimental drug; Women of reproductive age include premenopausal women and women within 1 year after menopause. Blood pregnancy test results for women of childbearing age must be negative within ≤7 days before the first trial drug administration.

Exclusion Criteria:

1. Tumors originating from nasopharyngeal, paranasal, nasal or salivary glands, thyroid or parathyroid lesions, skin, unknown primary squamous cell carcinoma or non-squamous histology (e.g., mucosal melanoma);
2. Peripheral neuropathy ≥ grade 2 (according to CTCAE v5.0);
3. Have received any of the following treatments:

   * Received intravenous antibiotic therapy within 7 days prior to initial dosing;
   * Investigational drugs that have received other clinical trials within 4 weeks prior to initial dosing;
   * have received live attenuated vaccine within 4 weeks prior to first administration, and are allowed to receive inactivated seasonal influenza vaccine or approved COVID-19 vaccine without live virus;
   * Received systemic immunostimulatory drugs (including but not limited to interferon, interleukin-2, etc.) within 4 weeks prior to initial administration;
   * Had major surgery (e.g., transabdominal, thoracic, etc., excluding diagnostic puncture, infusion device implantation, or digestive home implantation) within 4 weeks prior to initial dosing, or expected to require major surgery during the study period; Previous immunotherapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies (including ipilimumab) or any other antibody or drug that targets T-cell co-stimulation or immune checkpoint pathways;
4. A history of other primary malignancies within the past 3 years, excluding basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or cervical carcinoma in situ that has been completely and radically resected;
5. Clinically significant (i.e., active) cardiovascular disease: cerebrovascular accident/stroke/myocardial infarction, unstable angina, congestive heart failure (NYHA Class II and above), or severe arrhythmia requiring medication within the first 6 months of enrollment;
6. Evidence of active infection includes hepatitis B (HBsAg positive with HBV DNA≥2000 IU/ml, excluding hepatitis due to drugs or other causes), hepatitis C (HCV positive with anti-HCV antibody), hepatitis B (HCV positive with HBV DNA≥2000 IU/ mL), and hepatitis C (HCV positive with HBV DNA≥2000 IU/ mL). HCV RNA results greater than the lower limit of detection) or human immunodeficiency virus (HIV) infection; Uncontrolled active bacterial, other viral, fungal, rickettsial, or parasitic infections, unless treated and resolved prior to administration of the investigational drug;
7. Loss of more than 10% of body weight in the 4 weeks prior to the first dose (unless appropriate nutritional support measures are taken);
8. Active gastrointestinal bleeding, or bleeding requiring more than 2 red blood cell transfusions or 4 units of compressed red blood cell transfusions within the first 4 weeks;
9. Patients with a history of primary immunodeficiency or active autoimmune disease who were taking immunosuppressants or systemic hormone therapy (dose ≥10 mg/ day of prednisone or other equivalent hormone) and continued to use it within 2 weeks prior to enrollment; Attention: Patients with type I diabetes, stable hypothyroidism with hormone replacement therapy (including hypothyroidism due to autoimmune thyroid disease), psoriasis, vitiligo, or psoriasis that does not require systemic treatment may be enrolled with topical or inhaled corticosteroids, or short-term (≤7 days) corticosteroids for prevention or treatment of non-autoimmune diseases. And infrequent allergic diseases are excluded. ;
10. A history of grade 3 allergy to any component of MRG003, Ptrelizumab injection, and/or cisplatin injection;
11. Previous history of interstitial pneumonia, radiation pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.;
12. History of organ transplantation, including allogeneic peripheral stem cell or bone marrow transplantation. After careful evaluation, patients who received autologous hematopoietic stem cell transplantation (HSTC) ≥ 5 years ago and who have normal bone marrow function (independent of transfusion) may be considered for study participation;
13. Other conditions deemed unsuitable for participation in this clinical trial by the investigator, including but not limited to serious mental illness, central nervous disorder, substance abuse, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | After surgery (approximately 9-10 weeks after start of study treatment)
  Pathological complete response rate

SECONDARY OUTCOMES:
EFS EFS | 1 years
  Event free survival
ORR | 9-10 weeks
  Objective response rate
OS | 2 years
  Overall survival
Number of patients with Adverse Events (AEs) | Up to approximately 1 years
  79/5000 The incidence, severity and correlation of adverse events (AE), serious adverse events (SAE), immune-related adverse events (irAE), and laboratory index outliers were determined according to NCI-CTCAE v5.0 standards
Incidence of surgery-related AE/SAE (adverse events/serious adverse events) | 90 days
  Rate of delayed or canceled surgery, length of surgery, length of hospital stay, method of surgery, and incidence of surgery-related AE/SAE (adverse events/serious adverse events) within 90 days after surgery
Proportion of reduction in clinical stage after treatment | 9-10 weeks
  The proportion of clinical stage reduction after combination therapy in the target study population